CLINICAL TRIAL: NCT06658704
Title: Understanding Motivation Towards Exercise to Enhance Physical Activity on Prescription Adherence
Acronym: UMEPA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Andreas Hult, Associate Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2024-03415
Record Dates: First submitted 2024-10-18; First posted 2024-10-26 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Physical Inactivity
Keywords: Physical Inactivity; Exercise Referral Scheme; Physical activity on Prescription; Exercise intervention
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A two arm intervention study with allocation to usual care (Physical activity on Prescription) or usual care (Physical activity on Prescription) + an exercise intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise intervention (Experimental): Participants are prescribed a Physical activity on Prescription (PaP) which means that they will have a motivational interview with a physiotherapist regarding increased physical activity. The physiotherapist will then prescribe a individualized PaP with the goal to increase weekly physical activity that the participant are instructed to adhere to for the remainder of the study. A follow-up session is also included after 16 weeks. Participants are invited to a 16 week exercise intervention at a private fitness center after they have received their PaP. The exercise, including a variety of aerobic and resistance training, is performed in a group setting starting with one session per week for the first two weeks and then two sessions per week for week 3-16. Follow-up tests is also included after 6-, 12- and 24 months.
  Interventions: Behavioral: Supervised exercise in a group setting; Behavioral: Usual care (Physical activity on Prescription)
- Control (Active Comparator): Participants are prescribed a Physical activity on Prescription (PaP) which means that they will have a motivational interview with a physiotherapist regarding increased physical activity. The physiotherapist will then prescribe a individualized PaP with the goal to increase weekly physical activity that the participant are instructed to adhere to for the remainder of the study. A follow-up session is also included after 16 weeks. Follow-up tests is also included after 6-, 12- and 24 months.
  Interventions: Behavioral: Usual care (Physical activity on Prescription)

INTERVENTIONS:
Behavioral: Supervised exercise in a group setting — Participants are invited to a 16 week exercise intervention at a private fitness center after they have received their PaP. The exercise, including a variety of aerobic and resistance training, is performed in a group setting starting with one session per week for the first two weeks and then two sessions per week for week 3-16.
  Arms: Exercise intervention
Behavioral: Usual care (Physical activity on Prescription) — Participants are prescribed a Physical activity on Prescription (PaP) which means that they will have a motivational interview with a physiotherapist regarding increased physical activity. The physiotherapist will then prescribe a individualized PaP with the goal to increase weekly physical activity that the participant are instructed to adhere to for the remainder of the study. A follow-up session is also included after 16 weeks.

SUMMARY:
The goal of this clinical trial is to explore effectiveness on physical activity, function and psychometrics in relation to an exercise intervention in physically inactive middle-aged men and women. The main questions it aims to answer are:

* Is the exercise intervention effective in increasing physical activity, function and motivation towards exercise? Is there an intervention effect in physical activity, function and psychometrics at 6-, 12- and 24 months post baseline?
* Can barriers and facilitators towards increased physical activity be identified in the two groups of the study?

All participants will first receive standard care for physically inactive patients, i.e. Physical activity on Prescription (PaP), followed by allocation to an exercise intervention (EI) group or a control group. The EI group will be offered an additional exercise intervention for 16 weeks consisting of 1-2 training sessions per week of a combination of aerobic and resistance training at a private fitness centre. The control group will be asked to adhere to their PaP.

Researchers will assess physical activity, function and psychometrics in the two groups at 6-, 12- and 24 months to evaluate the intervention effect. Additionally, interviews with the participants in the control and EI groups will be performed in order to explore barriers and facilitators towards increased physical activity in formerly inactive patients.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive persons as defined as not meeting the current recommendations of at least 150 minutes of moderate to vigorous physical activity per week. This criterion is self-assessed by potential participants.
* Age 40-60 years

Exclusion Criteria:

* Physical disability that affects the ability to perform the exercise intervention.
* Heart failure or severe degenerative disease, e.g. malignant cancer, multiple sclerosis etc.
* Myocardial infarction or stroke during the last 12 months.
* Heart conditions including angina pectoris that is worsened with exercise.
* Neuromuscular, musculoskeletal, or rheumatic conditions that is worsened with exercise.
* Hypertension grade III, i.e. systolic blood pressure above 180 mmHg and/or diastolic blood pressure over 110 mmHg.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Self-reported exercise and physical activity | Baseline, 6-, 12- and 24 months
  One question regarding exercise and one question regarding every day physical activity in a typical week. The question regarding exercise comprises 6 answer alternatives ranging from 0 min to more than 120 min per week. The question regarding every day physical activity comprises 7 answer alternatives raging from 0 min to more than 300 min per week. The questions are produced by the Swedish National Board of Health and Welfare.

SECONDARY OUTCOMES:
Device measured physical activity level | Baseline, 6-, 12- and 24 months
  Device measured physical activity, measured with an accelerometer for 7 consecutive days. Raw data are then recalculated to minutes spent in light, moderate and vigouros physical acticity intensity zones.
Daily step count | Baseline, 6-, 12- and 24 months
  Data from device measured physical activity, measured with an accelerometer for 7 consecutive days, are used to collect daily step counts.
Cardio-respiratory capacity | Baseline, 6-, 12- and 24 months
  Ekblom-Bak cycle ergometer test will be used to assess cardio-respiratory fitness.
Upper limb strength | Baseline, 6-, 12- and 24 months
  Hand grip strength of the non dominant hand is measured with a hand dynamometer to the nearest kg. Three consecutive trials is performed in a seated position with the elbow held at a 90 degree angle and the highest value is recorded. A higher value indicate higher upper limb strength.
Lower limb muscle strength | Baseline, 6-, 12- and 24 months
  Five repetition sit to stand test. From a seated position, the participant is instructed to stand up and then sit down again for a total of five times. The total time of five repetition sit to stand cycles is then recorded in seconds with a stopwatch. A lower total time indicate higher lower limb muscle strength.
Motivational stages of self-determination for exercise | Baseline, 6-, 12- and 24 months
  Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2) will be used. The questionnaire contains 19 questions, belonging to one of the five categories Amotivation, External regulation, Introjected regulation, Identified regulation and Intrinsic regulation. The scale assesses where a person is on the continuum of self-determination in where higher, positive scores indicate greater relative autonomy; lower, negative scores indicate more controlled regulation.
Confidence in one's own ability to exercise | Baseline, 6-, 12- and 24 months
  The Swedish Exercise Self-Efficacy Scale (ESES-S) will be used. The questionnaire comprises 10 questions on exercise self-efficacy, each with four answer alternatives. The composite score ranges from 10 to 40 and a higher score indicate a higher precised self-efficacy towards exercise.
Basic psychological needs connected to physical activity satisfaction | Baseline, 6-, 12- and 24 months
  The Basic Psychological Needs in Exercise Scale (BPNES) will be used. This questionnaire contains 12 questions related to one of three basic psychological needs; Autonomy, Competence and Relatedness in the exercise domain. Answers are given on a five point Likert scale and results are presented for the individual needs and as a collective, global need. The maximal score for each question is 5 and the minimal score is 1. Mean values for each need is presented together with a mean score of all 12 questions. A higher score indicate a higher need fulfillment.
Health related quality of life | Baseline, 6-, 12- and 24 months
  RAND-36 health survey will be used (RAND is not an acronym but the name of a research corporation). The RAND-36 survey contains 36 questions belonging to eight health concepts that can be further categorized into two summary scores; physical and mental health. The answers from the survey is re-coded into points in where higher points indicate better perceived health. The points, ranging from 0 to 100, are then presented for the different concepts, the two summary scores and the overall score for the 36 questions.

OTHER OUTCOMES:
Exploring barriers and facilitators towards physical activity | 12- and/or 24 months
  Semi-structured qualitative individual interviews will be conducted in both groups where barriers and facilitators towards physical activity will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hult, PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No
Sharing of individual data is not in accordance with the ethical permission granted from the Swedish ethics review authority.